CLINICAL TRIAL: NCT05392530
Title: A Single-center, Open-label, Single-dose, Randomized, 3-way Crossover Phase 1 Study in Healthy Adult Participants to Assess the Relative Oral Bioavailability of Macitentan 75 mg as Two Different Test Formulations Compared to the Reference Formulation
Brief Title: A Study of Two Different Test Formulations Compared to the Reference Formulation of Macitentan in Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Actelion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: CR109202; 2022-000275-39 (EudraCT Number); 67896062PAH1012 (Other: Actelion)
Record Dates: First submitted 2022-05-23; First posted 2022-05-26 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Healthy
MeSH Terms: interventions — macitentan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Treatment Sequence ABC (Experimental): Participants will receive single oral dose of final marketing image (FMI) candidate #1 of macitentan (Treatment A [test]) under fed condition in Treatment Period 1, followed by single oral dose of FMI candidate #2 of macitentan (Treatment B [test]) under fed conditions in Treatment Period 2, and then single oral dose of the reference formulation of macitentan (Treatment C) under fed conditions in Treatment Period 3. The study intervention administrations will be separated by at least 14 days to allow adequate washout duration following the single doses.
  Interventions: Drug: Macitentan
- Treatment Sequence BCA (Experimental): Participants will receive Treatment B in Treatment Period 1 followed by Treatment C in Treatment Period 2, and then Treatment A in Treatment Period 3 on Day 1. The study intervention administrations will be separated by at least 14 days to allow adequate washout duration following the single doses.
  Interventions: Drug: Macitentan
- Treatment Sequence CAB (Experimental): Participants will receive Treatment C in Treatment Period 1 followed by Treatment A in Treatment Period 2, and then Treatment B in Treatment Period 3 on Day 1. The study intervention administrations will be separated by at least 14 days to allow adequate washout duration following the single doses.
  Interventions: Drug: Macitentan
- Treatment Sequence ACB (Experimental): Participants will receive Treatment A in Treatment Period 1 followed by Treatment C in Treatment Period 2, and then Treatment B in Treatment Period 3 on Day 1. The study intervention administrations will be separated by at least 14 days to allow adequate washout duration following the single doses.
  Interventions: Drug: Macitentan
- Treatment Sequence CBA (Experimental): Participants will receive Treatment C in Treatment Period 1 followed by Treatment B in Treatment Period 2, and then Treatment A in Treatment Period 3 on Day 1. The study intervention administrations will be separated by at least 14 days to allow adequate washout duration following the single doses.
  Interventions: Drug: Macitentan
- Treatment Sequence BAC (Experimental): Participants will receive Treatment B in Treatment Period 1 followed by Treatment A in treatment period 2, and then Treatment C in Treatment Period 3 on Day 1. The study intervention administrations will be separated by at least 14 days to allow adequate washout duration following the single doses.
  Interventions: Drug: Macitentan

INTERVENTIONS:
Drug: Macitentan — Macitentan film coated tablets will be administered orally as per assigned treatment sequence.
  Other Names: Opsumit

SUMMARY:
The purpose of this study is to assess the rate and extent of absorption of a single oral dose of macitentan given as 2 test formulations compared to the reference formulation under fed conditions in healthy adult participants.

ELIGIBILITY:
Inclusion Criteria:

* Healthy on the basis of physical examination and medical and surgical history, performed at screening. If there are abnormalities, the participant may be included only if the investigator judges the abnormalities to be not clinically significant. This determination must be recorded in the participant's source documents and initialed by the investigator
* Systolic blood pressure (SBP) between 100 and 145 millimeters of mercury (mmHg) (inclusive), diastolic blood pressure (DBP) between 50 and 90 mmHg (inclusive), and pulse rate between 45 and 90 beats per minute (inclusive), within 3 minutes after standing up and after the participant is supine for at least 5 minutes, at screening
* Twelve-lead electrocardiogram (ECG) without clinically relevant abnormalities, at the discretion of the investigator, measured after the participant is supine for at least 5 minutes, at screening
* Body weight not less than 50 kilograms (Kg) and body mass index (BMI; weight/height^2) within the range 18.5 -30 kg per meter square (kg/m^2) (inclusive)at screening
* All women must have a negative highly sensitive serum (beta-human chorionic gonadotropin [beta-hCG]) pregnancy test at screening and a negative urine pregnancy test on Day -1 of the first treatment period

Exclusion Criteria:

* Known allergies, hypersensitivity, or intolerance to any active substance or drugs of the same class, or any excipient of the drug formulation(s)
* History or clinical evidence of any disease and/or existence of any surgical or medical condition which might interfere with the absorption, distribution, metabolism, or excretion of the study intervention(s) (appendectomy and herniotomy allowed, cholecystectomy not allowed)
* A history of repeated fainting due to cardiac cause, collapse, syncope, orthostatic hypotension, or vasovagal reactions
* Female participant who is breastfeeding at screening and plans to breastfeed throughout the study
* Any condition for which, in the opinion of the investigator, participation would not be in the best interest of the participant (example, compromise the well-being) or that could prevent, limit, or confound the protocol-specified assessments

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2022-05-25 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2022-09-14 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Analyte Concentration (Cmax) of Macitentan | Predose, up to 336 hours post dose (up to Day 15)
  Cmax is defined as maximum observed plasma analyte concentration of macitentan.
Area Under the Plasma Analyte Concentration-time Curve from Time Zero to Time of the Last Quantifiable Concentration of Macitentan (AUC[0-last]) | Predose, up to 336 hours post dose (up to Day 15)
  AUC(0-last) is defined as area under the plasma analyte concentration-time curve of macitentan from time zero to time of the last quantifiable (non-below quantification limit [BQL]) concentration.
Area Under the Plasma Analyte Concentration-time Curve from Time Zero to Infinite Time (AUC[0-infinity]) of Macitentan | Predose, up to 336 hours post dose (up to Day 15)
  AUC(0-infinity) is defined as area under the plasma analyte concentration-time curve of macitentan from time zero to infinite time.

SECONDARY OUTCOMES:
Actual Sampling Time to Reach the Maximum Observed Plasma Analyte Concentration (Tmax) of Macitentan and its Metabolite Aprocitentan | Predose, up to 336 hours post dose (up to Day 15)
  Tmax is defined as actual sampling time to reach the maximum observed plasma analyte concentration of macitentan and its metabolite aprocitentan.
Last Observed Measurable Plasma Analyte Concentration (Clast) of Macitentan and its Metabolite Aprocitentan | Predose, up to 336 hours post dose (up to Day 15)
  Clast is defined as last observed measurable plasma analyte concentration of macitentan and its metabolite aprocitentan.
Area Under the Plasma Analyte Concentration-time Curve of Macitentan and its Metabolite Aprocitentan from Time Zero to 72 Hours Post dose (AUC[0-72 Hours]) | Predose, up to 336 hours post dose (up to Day 15)
  AUC(0-72 hours) is defined as area under the plasma analyte concentration-time curve of macitentan and its metabolite aprocitentan from time zero to 72 hours post dose, calculated by linear-linear trapezoidal summation.
Apparent Terminal Elimination Half-life (t1/2) of Macitentan and its Metabolite Aprocitentan | Predose, up to 336 hours post dose (up to Day 15)
  t1/2 is defined as apparent terminal elimination half-life of macitentan and its metabolite aprocitentan.
Apparent Terminal Elimination Rate Constant (Lambda[z]) of Macitentan and its Metabolite Aprocitentan | Predose, up to 336 hours post dose (up to Day 15)
  Lambda(z) is defined as apparent terminal elimination rate constant of macitentan and its metabolite aprocitentan, estimated by linear regression using the terminal log-linear phase of the log transformed concentration versus time curve.
Total Apparent Oral Clearance (CL/F) of Macitentan | Predose, up to 336 hours post dose (up to Day 15)
  CL/F of macitentan is defined as total apparent oral clearance, calculated as dose/AUC (0-infinity).
Apparent Volume of Distribution (Vdz/F) of Macitentan | Predose, up to 336 hours post dose (up to Day 15)
  Vdz/F of macitentan is defined as apparent volume of distribution, calculated as dose/(Lambda[z]*AUC [0-infinity]).
Maximum Observed Plasma Analyte Concentration (Cmax) of Aprocitentan | Predose, up to 336 hours post dose (up to Day 15)
  Cmax is defined as maximum observed plasma analyte concentration of metabolite aprocitentan.
Area Under the Plasma Analyte Concentration-Time Curve from Time Zero to Time of the Last Quantifiable Concentration of Aprocitentan (AUC[0-last]) | Predose, up to 336 hours post dose (up to Day 15)
  AUC(0-last) of metabolite Aprocitentan is defined as area under the plasma analyte concentration-time curve from time zero to time of the last quantifiable (BQL) concentration, calculated by linear-linear trapezoidal summation.
Area Under the Plasma Analyte Concentration-Time Curve of Aprocitentan from Time Zero to Infinity (AUC[0-infinity]) | Predose, up to 336 hours post dose (up to Day 15)
  AUC(0-infinity) is defined as area under the plasma analyte concentration-time curve of metabolite aprocitentan from time zero to infinite time.
Number of Participants with Serious Adverse Events (SAEs) | Up to 13 weeks
  Number of Participants with Serious Adverse Events (SAEs) will be reported SAE is any untoward medical occurrence that at any dose may results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, is a suspected transmission of any infectious agent via a medicinal product.
Number of Participants with Adverse Events (AEs) | Up to 13 weeks
  Number of participants with AEs will be reported. An AE is any untoward medical occurrence in a clinical study participant administered a pharmaceutical (investigational or non investigational) product.
Number of Participants with Abnormalities in Physical Examination | Up to Day 15
  Number of participants with abnormalities in physical examination (including general appearance, respiratory, neurological, eyes, ear/nose/throat, thyroid, cardiovascular, abdominal/gastrointestinal, hepatic, musculoskeletal, and dermatologic) will be reported.
Number of Participants with Abnormalities in Vital Signs | Up to Day 15
  Number of participants with abnormalities in vital signs (including temperature [tympanic], pulse rate, and blood pressure) will be reported.
Number of Participants with Abnormalities in Electrocardiograms (ECGs) | Up to Day 15
  Number of participants with abnormalities in ECGs will be reported.
Number of Participants with Abnormalities in Clinical Laboratory Tests | Up to Day 15
  Number of participants with abnormalities in clinical laboratory tests (including serum chemistry, hematology, and urinalysis) will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Actelion Clinical Trial, Study Director — Actelion
Locations (1):
- SGS Belgium NV, Edegem, Belgium

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency